CLINICAL TRIAL: NCT07245056
Title: Evaluation of the Fetal Fornix and Hippocampus in Pregnant Women With Early-Onset Preeclampsia
Brief Title: Fetal Fornix and Hippocampus in Pregnant Women With Early-Onset Preeclampsia
Acronym: FHC-EOPE
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Ankara Etlik City Hospital (Other Government)
Responsible Party: Principal Investigator, Seyit Ahmet Erol, Associate Professor, MD, Ankara Etlik City Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: AEŞH-BADEK2-2025-551
Record Dates: First submitted 2025-11-15; First posted 2025-11-24 (Actual); Last update posted 2025-12-23 (Actual); Status verified 2025-12

CONDITIONS: Pre-Eclampsia; Hippocampus
Keywords: fetal brain; fornix; hippocampus; early-onset preeclampsia
MeSH Terms: conditions — Pre-Eclampsia | interventions — eosinylphosphatidylethanolamine; Control Groups

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- One arm (fetal FHC measurements for EOPE and control groups) (Other): One arm for fetal fornix and hippocampus complex (FHC) measurements on early-onset preeclampsia (EOPE) and control groups
  Interventions: Other: FHC dimensions in EOPE and control groups

INTERVENTIONS:
Other: FHC dimensions in EOPE and control groups — Fetal fornix and hippocampus complex (FHC) dimension changes on EOPE and control groups

SUMMARY:
Since early-onset preeclampsia (EOPE) is commonly associated with inadequate placentation, placental insufficiency, chronic fetal hypoxia, oxidative stress, and heightened inflammation, these pathological processes may adversely affect hippocampal neuronal development and maturation of axonal pathways such as the fornix. These mechanisms support our hypothesis that fetal fornix and hippocampus dimensions may be reduced in pregnancies complicated by EOPE, forming the scientific basis of our study.

Previous research has suggested a potential link between preeclampsia (PE) and altered neurocognitive development. However, no studies to date have specifically evaluated the relationship between EOPE and fetal fornix or hippocampus dimensions. Therefore, the objective of our study is to assess fetal fornix and hippocampus measurements in pregnant women with early-onset preeclampsia compared with healthy controls.

DETAILED DESCRIPTION:
Hypertensive disorders complicate approximately 5-10% of all pregnancies and account for nearly 16% of maternal mortality. Preeclampsia (PE) occurs in 4-5% of pregnancies, and in the United States, preeclampsia or eclampsia contributed to 7.4% of the 2,009 pregnancy-related maternal deaths reported between 2011 and 2013. Preeclampsia is defined by new-onset hypertension and proteinuria, or new-onset hypertension with or without proteinuria, accompanied by evidence of significant end-organ dysfunction. It is a progressive, multisystem disorder that generally develops after 20 weeks of gestation or during the postpartum period.

Preeclampsia is also considered a pregnancy-specific syndrome capable of affecting every organ system. Because of its significant maternal and perinatal morbidity and mortality, PE represents a major public health concern. The condition is commonly described as a two-stage disease. Stage 1 (placental syndrome) is characterized by early placental ischemia/reperfusion, oxidative stress, and the release of toxic factors, primarily due to abnormal endovascular trophoblastic remodeling, primigravidity, trophoblast load, genetic predisposition, and maternal immunologic maladaptation. Stage 2 (maternal syndrome) represents the clinical phase, driven by an exaggerated maternal systemic inflammatory response and endothelial dysfunction. Maternal genetic susceptibility and underlying vascular disease may further contribute.

Overall, the etiopathogenesis of PE involves abnormal trophoblastic invasion, maternal-fetal immunologic incompatibility, maladaptation to normal cardiovascular and inflammatory changes of pregnancy, systemic vascular dysfunction, genetic influences, and epigenetic mechanisms. Approximately 90% of preeclampsia cases occur in the late-preterm (34-37 weeks), term, or postpartum period and generally have more favorable outcomes. However, severe morbidity and mortality may still occur. The remaining 10% of cases present as early-onset preeclampsia (EOPE, <34 weeks), in which abnormal placentation and defective trophoblastic invasion are more pronounced and closely correlate with disease severity. EOPE carries a markedly higher risk of serious perinatal complications, largely due to its strong association with preterm delivery. Consequently, the study of EOPE remains clinically important.

The hippocampus is a seahorse-shaped structure located within the medial temporal lobe, protruding laterally toward the temporal horn of the lateral ventricle. It plays essential roles in memory processing (dorsal hippocampus) and regulation of stress responses (ventral hippocampus). Fetal hippocampal development involves progressive inward folding of the dentate gyrus, cornu ammonis, subiculum, and parahippocampal gyrus around the shrinking hippocampal sulcus.

Experimental studies have demonstrated that adverse maternal conditions may affect hippocampal development. In rodent models, uncontrolled maternal diabetes reduces hippocampal volume and neuronal density during early postnatal life, leading to delayed development and motor, behavioral, and cognitive deficits in offspring. In an experimental preeclampsia model induced with a cholesterol-based diet, hippocampal arteriolar vasoreactivity to neurovascular coupling mediators was impaired, resulting in deficits in long-term-but not spatial-memory. These findings may parallel long-term cardiovascular and neurocognitive outcomes observed in women with a history of preeclampsia and eclampsia. Persistent endothelial and vascular smooth muscle dysfunction in hippocampal vessels may contribute to disrupted hippocampal networks and early cognitive impairment.

Clinical and experimental data also suggest that children born to preeclamptic mothers have higher rates of neurodevelopmental disorders, including cognitive impairments, autism spectrum disorder, depressive disorders, attention-deficit/hyperactivity disorder, and cerebral palsy. Reported neuronal abnormalities include impaired neurogenesis, reduced neuronal integrity, accumulation of cellular debris, decreased synaptogenesis and myelination, and abnormal neurite outgrowth, potentially mediated by microglial activation, inflammation, and reduced angiogenesis.

Since EOPE is frequently associated with inadequate placentation, placental insufficiency, chronic fetal hypoxia, oxidative stress, and inflammation, these pathophysiologic processes may interfere with fetal hippocampal neuronal development and maturation of the fornix. These mechanisms support our hypothesis that fetal fornix and hippocampus dimensions may be reduced in EOPE.

Ultrasonographic literature on fetal hippocampal imaging is limited. Gindes et al. demonstrated that the fetal hippocampus and fornix can be identified as a C-shaped structure on sagittal three-dimensional (3D) ultrasound. Toprak et al. reported that the fetal fornix and hippocampus can be rapidly visualized using two-dimensional (2D) ultrasound during midtrimester anomaly screening. Sahin et al. confirmed that the bilateral fornix-hippocampus complex can be visualized between 18 and 36 weeks of gestation and proposed sonographic reference values.

Research Hypothesis:

Is there a difference in fetal fornix and hippocampus dimensions in pregnancies complicated by early-onset preeclampsia compared with healthy controls? Our primary hypothesis is that fetal fornix and hippocampus dimensions are reduced in EOPE.

Expected Benefits:

By assessing the relationship between fetal fornix and hippocampus size and EOPE, and evaluating potential associations with pregnancy prognosis and complications, this study may contribute to improved understanding and management of the condition and support future prospective research. The study poses no risk to pregnant women or fetuses.

The study will enroll 42 pregnant women diagnosed with EOPE (aged 18-45 years, 20-34 weeks of gestation) presenting to the Perinatology Clinic of Ankara Etlik City Hospital, along with 42 healthy controls. Sample size calculation using G*Power 3.1.9.7 indicated that a minimum of 84 participants would provide 95% statistical power (effect size d = 0.8, α = 0.05, 1-β = 0.95). Participants will be included after informed consent is obtained, and confidentiality will be ensured.

Demographic and routinely collected clinical data-including age, gestational age, height, weight, BMI, weight gain, gravidity, parity, obstetric history, comorbidities, medications, prior surgeries, tobacco and alcohol use-will be recorded. Routine laboratory parameters and ultrasonographic measurements (biometry, amniotic fluid index, umbilical artery Doppler systolic/diastolic (S/D) ratio and pulsatility index (PI), middle cerebral artery Doppler peak systolic velocity (PSV) and PI, uterine artery Doppler PI, cerebroplacental ratio (CPR), and cerebro-placento-uterine ratio (CPUR)) will also be obtained.

For this study, fetal fornix and hippocampus dimensions will be measured by 2D ultrasound in both EOPE and control groups using standard clinic equipment. All findings will be compiled into a detailed report including statistical analyses, comparisons between groups, and evaluation of the relationship between EOPE and fetal fornix/hippocampus measurements.

ELIGIBILITY:
Inclusion Criteria:

* Women aged 18-45 years
* Gestational age between 20 and 34 weeks
* Diagnosis of early-onset preeclampsia (EOPE)
* Singleton pregnancy

Exclusion Criteria:

* Multiple pregnancies
* Presence of chronic or significant comorbid conditions other than maternal early-onset preeclampsia, including: Chronic, mental, or physical illnesses, severe renal, hepatic, or gastrointestinal acute or chronic inflammatory diseases, hyperthyroidism or hypothyroidism, chronic hypertension, type 1 or type 2 diabetes mellitus, history of polycystic ovary syndrome (PCOS), history of malignancy
* Fetal congenital or chromosomal anomalies
* Chronic medication use
* Tobacco or alcohol use during pregnancy
* Maternal late-onset preeclampsia (≥34 weeks gestation)

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Pregnant women
Enrollment: 84 (Estimated)
Dates: Start 2025-12-01 (Actual); Primary Completion 2026-07-01 (Estimated); Study Completion 2026-08-01 (Estimated)

PRIMARY OUTCOMES:
Fetal fornix-hippocampus complex (FHC) dimensions (mm) | Until completion of participant recruitment (approximately 7 months).
  Measurement of fetal fornix-hippocampus complex (FHC) length and hippocampus height using two-dimensional ultrasonography (2D-US) in pregnancies complicated by early-onset preeclampsia (EOPE) compared with healthy controls.
  Unit of Measure: Millimeters (mm) Measurement Tool: Two-dimensional ultrasonography (2D-US)

SECONDARY OUTCOMES:
Correlation between fetal FHC and hippocampus height measurements and composite adverse perinatal outcomes | Until completion of participant recruitment (approximately 7 months).
  Assessment of the correlation between fetal Fornix-Hippocampus Complex (FHC) and hippocampus height measurements obtained by 2D ultrasonography and composite adverse perinatal outcomes, specifically preterm birth <34 weeks (reported as both absolute number and percentage), fetal growth restriction (FGR), NICU admission, and low Apgar scores.
  Unit of Measure: Correlation coefficient (r)
  Measurement Tools:
  * FHC and hippocampus height measurements by 2D ultrasonography
  * Perinatal outcome data obtained at delivery

CONTACTS AND LOCATIONS:
Overall Officials: Seyit A Erol, MD, Principal Investigator — Ankara Etlik City Hospital
Locations (1):
- Ankara Etlik City Hospital, Ankara, Yenimahalle, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No
The data that support the findings of this study are available from the central contact person, upon reasonable request.

REFERENCES:
- [Background] Zhang H, Lin J, Zhao H. Impacts of Maternal Preeclampsia Exposure on Offspring Neuronal Development: Recent Insights and Interventional Approaches. Int J Mol Sci. 2024 Oct 15;25(20):11062. doi: 10.3390/ijms252011062. PMID 39456854
- [Background] Johnson AC, Li Z, Orfila JE, Herson PS, Cipolla MJ. Hippocampal network dysfunction as a mechanism of early-onset dementia after preeclampsia and eclampsia. Prog Neurobiol. 2021 Apr;199:101938. doi: 10.1016/j.pneurobio.2020.101938. Epub 2020 Oct 29. PMID 33130230
- [Background] Johnson AC, Tremble SM, Cipolla MJ. Experimental Preeclampsia Causes Long-Lasting Hippocampal Vascular Dysfunction and Memory Impairment. Front Physiol. 2022 May 9;13:889918. doi: 10.3389/fphys.2022.889918. eCollection 2022. PMID 35615682
- [Background] Sadeghi A, Asghari H, Hami J, Mohasel Roodi M, Mostafaee H, Karimipour M, Namavar M, Idoon F. Volumetric investigation of the hippocampus in rat offspring due to diabetes in pregnancy-A stereological study. J Chem Neuroanat. 2019 Nov;101:101669. doi: 10.1016/j.jchemneu.2019.101669. Epub 2019 Aug 20. PMID 31442582
- [Result] Arica G, Davutoglu EA, Buldum D, Kucuksuleymanoglu D, Najmeddin S, Madazli R. Fetal Fornix-Hippocampus Complex and Hippocampus Height Measurements Between 18 and 24 Weeks of Gestation and the Effect of Maternal Iron Deficiency Anemia. J Clin Ultrasound. 2025 Jul-Aug;53(6):1288-1295. doi: 10.1002/jcu.24008. Epub 2025 Apr 16. PMID 40237113
- [Result] Gindes L, Weissmann-Brenner A, Weisz B, Zajicek M, Geffen KT, Achiron R. Identification of the fetal hippocampus and fornix and role of 3-dimensional sonography. J Ultrasound Med. 2011 Dec;30(12):1613-8. doi: 10.7863/jum.2011.30.12.1613. PMID 22123994
- [Result] Sahin NE, Alici Davutoglu E, Arica G, Madazli R. Identification of bilateral fornix and hippocampus in fetuses between 18-36 gestational weeks and establishment of nomograms using ultrasonography. Arch Gynecol Obstet. 2025 Aug;312(2):627-634. doi: 10.1007/s00404-025-08061-z. Epub 2025 May 23. PMID 40407880
- [Result] Toprak E, Sayal HB. Ultrasonographic imaging of the fetal hippocampus. Arch Gynecol Obstet. 2024 May;309(5):1943-1949. doi: 10.1007/s00404-023-07093-7. Epub 2023 Jun 9. PMID 37294452